CLINICAL TRIAL: NCT02706275
Title: Pilot Randomized Trial of External Warming in Critically Ill Adult Septic Patients
Brief Title: Pilot Trial of External Warming in Septic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201512121
Record Dates: First submitted 2016-03-01; First posted 2016-03-11 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Warming Group (Experimental): External warming via forced air warming
  Interventions: Other: External warming
- Control Group (No Intervention): Standard of care body temperature management

INTERVENTIONS:
Other: External warming — External warming via forced air warming to a goal body temperature 1.5°C greater than the baseline minimum temperature (within previous 24 hours) for 48 hours
  Arms: Warming Group

SUMMARY:
The purpose of this study is to determine whether externally warming critically ill afebrile adult septic patients will improve indices of immune function and/or clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a surgical or medical intensive care unit
* Age greater than 18 years
* Diagnosis of sepsis within 24 hours of enrollment
* Requirement for mechanical ventilation with expected duration of mechanical ventilation > 48 hours
* Goal Richmond Agitation Sedation Scale (RASS) < 0
* Maximum baseline temperature (within previous 24 hours) < 38.3°C

Exclusion Criteria:

* Treatment with chemotherapy within 6 months of enrollment
* Treatment with corticosteroids at a dose > 300 mg/day hydrocortisone (or equivalent)
* History of solid organ transplant on any immunosuppression medication
* History of immunological disease
* History of chronic infection with hepatitis B or C virus
* History of acute stroke, acute coronary syndrome, or severe head injury requiring osmotic therapy within 7 days prior to enrollment
* History of multiple sclerosis
* Contraindications to both bladder or esophageal core temperature monitors or to forced air warming blankets
* Moribund status
* Sepsis without source control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-05-12 (Actual); Study Completion 2019-05-12 (Actual)

PRIMARY OUTCOMES:
Monocyte human leukocyte antigen (mHLA-DR) expression | 48 hours hours following the start of the intervention period

SECONDARY OUTCOMES:
Interferon (IFN)-gamma production | 48 hours following the start of the intervention period
Number of patients who acquire nosocomial infections | 30 days after diagnosis of sepsis
  Number of patients who develop a nosocomial infection (defined as a new infection diagnosed greater than 48 hours after the original sepsis diagnosis) within 30 days of the sepsis diagnosis
Mortality | 28 days
Number of patients in whom the intervention is stopped early secondary to hemodynamic changes related to the intervention | Through study completion, 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Drewry AM, Mohr NM, Ablordeppey EA, Dalton CM, Doctor RJ, Fuller BM, Kollef MH, Hotchkiss RS. Therapeutic Hyperthermia Is Associated With Improved Survival in Afebrile Critically Ill Patients With Sepsis: A Pilot Randomized Trial. Crit Care Med. 2022 Jun 1;50(6):924-934. doi: 10.1097/CCM.0000000000005470. Epub 2022 Feb 7. PMID 35120040